CLINICAL TRIAL: NCT01719471
Title: fMRI of Stress in Smoking Behavior
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0805003898; RL1AA017539 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Smokers: Nicotine dependent individuals otherwise medically healthy
- Healthy: Medically healthy individuals who do not smoke

SUMMARY:
To examine the influence of current daily tobacco smoking on brain activation during stress, tobacco cue, and neutral relaxing conditions

DETAILED DESCRIPTION:
Subjects will participate in an fMRI session to examine changes in frontal and limbic brain regions with tobacco cues, stress and neutral/relaxing imagery. During each fMRI session subjects will participate in six imagery trials: 2 different neutral/relaxing, 2 different stress and 2 different tobacco cue scripts.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-50 years inclusive;
2. able to read and write English;
3. for women, being in follicular phase of menstrual cycle;

5) Tobacco dependent sample: smokes 10 or more cigarettes daily for the past year; Non-smokers, no tobacco consumption for more than one year and never having used tobacco daily.

Exclusion Criteria:

1. any major neurological illness or injury and any current or prior clinically significant mental health (including PTSD) or substance use disorder (with possible exception of nicotine dependence) as determined by SCID interview;
2. use of any psychoactive medication within past four weeks;
3. any significant unstable medical condition such as asthma or heart disease for which increased cardiovascular reactivity during stress challenge might constitute a significant risk;
4. IQ<70 based on past intelligence testing;
5. any metal in body that would pose a risk with MRI; and
6. claustrophobia that would interfere with MRI;
7. alcohol and drug use in the 72 hours prior to scanning, with the exception of tobacco;
8. pregnancy for women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 tobacco dependent and 30 matched healthy controls who have never smoked will be recruited for this study
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
No outcome measures for this study, this is an imaging study only | Upon study completion

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States